CLINICAL TRIAL: NCT03225612
Title: Safety and Performance of the Trialign Percutaneous Tricuspid Valve Annuloplasty System (PTVAS) for Symptomatic Chronic Functional Tricuspid Regurgitation
Brief Title: Safety and Performance of the Trialign Percutaneous Tricuspid Valve Annuloplasty System (PTVAS)
Acronym: SCOUT-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mitralign, Inc. (Industry)
Collaborators: Genae (Industry); Regulatory and Clinical Research Institute Inc (Other); CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLPR-011
Record Dates: First submitted 2017-06-14; First posted 2017-07-21 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Chronic Symptomatic Functional Tricuspid Regurgitation; Tricuspid Valve Insufficiency; Heart Valve Disease
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Open Label (Experimental): Non-randomized, open label clinical study that intends to treat up to 60 subjects with the Mitralign Percutaneous Tricuspid Valve Annuloplasty System (PTVAS) using standard of care techniques and services that are typically used for structural heart procedures.
  Interventions: Device: Mitralign Percutaneous Tricuspid Valve Annuloplasty System (PTVAS)

INTERVENTIONS:
Device: Mitralign Percutaneous Tricuspid Valve Annuloplasty System (PTVAS) — Mitralign Percutaneous Tricuspid Valve Annuloplasty System (PTVAS) is delivered by a percutaneous transcatheter procedure. The Trialign PTVAS procedure utilizes catheters and wires to deliver up to two sets of pledgeted sutures across the tricuspid annulus near the septal/posterior and the posterior/anterior commissures. Each set of implants is pulled together to plicate the posterior tricuspid annulus.

SUMMARY:
The purpose of this study is to assess the safety and performance of the Trialign System for the treatment of symptomatic chronic functional tricuspid regurgitation (FTR) in patients with a minimum of moderate tricuspid regurgitation.

The procedure will be performed with the PTVAS device using a non-surgical percutaneous approach to tricuspid valve repair in patients who have FTR with a minimum of moderate tricuspid regurgitation.

DETAILED DESCRIPTION:
A prospective, single-arm, multi-center study, enrolling symptomatic patients with chronic functional tricuspid regurgitation. The study will include up to 60 subjects from up to 15 sites in Europe and the United States. Follow-up evaluations will be conducted through 5 years post implantation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic functional tricuspid regurgitation (FTR) with a minimum of moderate tricuspid regurgitation;
* ≥18 and ≤85 years old;
* NYHA II, III, or ambulatory IV;
* Symptomatic despite Guideline Directed medical Therapy (GDMT), at minimum, patient on diuretic use;
* patient is at high risk for open heart valve surgery
* LVEF ≥35%
* Tricuspid valve annular diameter ≤55 mm (or 29 mm/m^2)

Exclusion Criteria:

* Pregnant or lactating female;
* Severe uncontrolled hypertension (SBP ≥ 180 mmHg and/or DBP ≥ 110 mmHg);
* Previous tricuspid valve repair or replacement;
* Severe coronary artery disease;
* MI or known unstable angina within the 30-days prior to the index procedure;
* Any PCI within 30 days prior to the index procedure or planned 3 months post the index procedure;
* Chronic oral steroid use (≥6 months);
* Life expectancy of less than 12-months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of all-cause mortality at 30 days. | 30-days
  Incidence of all-cause mortality at 30 days.

SECONDARY OUTCOMES:
Technical success | 30 Days
  Technical success, defined as freedom from death at 30 days with:
  * successful access, delivery and retrieval of the device delivery system;
  * deployment and correct positioning of the intended device(s) which is maintained and;
  * no need for additional unplanned or emergency surgery or re-intervention related to the device or access procedure
Echocardiographic variable: tenting height (maximum, any view) | Change from Baseline at 30 days
  Echocardiographic variables assessed by the Echocardiographic Core Lab at baseline and 30-days reflecting the severity of tricuspid pathology and the response to the Trialign device
Echocardiographic variable: tenting area (maximum, any view) | Change from Baseline at 30 days
  Echocardiographic variable assessed by the Echocardiographic Core Lab at baseline and 30-days reflecting the severity of tricuspid pathology and the response to the Trialign device
Echocardiographic variable: Quantification of tricuspid valve and annular area (maximum, any view) | Change from Baseline at 30 days
  Echocardiographic variable assessed by the Echocardiographic Core Lab at baseline and 30-days reflecting the severity of tricuspid pathology and the response to the Trialign device
Tricuspid regurgitation as determined by echocardiographic methods | Change from Baseline at 30 days
  As measured by the PISA method and the Quantitative Flow method
Percent tricuspid regurgitation from baseline to 30-days | Change from Baseline at 30 days
  Percent tricuspid regurgitation from baseline to 30-days
Adverse Events | Up to 60 months post procedure
  Rate of adverse events, including serious adverse events
New York Heart Association (NYHA) classification | Change from Baseline at discharge and then 1, 3, 6, 12, 24, 36, 48 and 60 months post procedure
  Change in New York Heart Association (NYHA) classification
Six-Minute Walk Test (6MWT) | Change from Baseline at discharge and then 1, 3, 6, 12, 24, 36, 48 and 60 months post procedure
  Change in the Six-Minute Walk Test (6MWT)
Minnesota Living with Heart Failure Questionnaire (MLWHF) | Change from Baseline at discharge and then 1, 3, 6, 12, 24, 36, 48 and 60 months post procedure
  Score on the Minnesota Living with Heart Failure Questionnaire (MLWHF)
EuroQol Five Dimensions Questionnaire (EQ-5D) | Change from Baseline at discharge and then 1, 3, 6, 12, 24, 36, 48 and 60 months post procedure
  Score on the EuroQol Five Dimensions Questionnaire (EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med Joachim Schofer, Principal Investigator — Medizinisches Versorgungszentrum Prof. Mathey, Prof. Schofer GmbH
Locations (11):
- Germany (6):
  - Vivantes Klinikum Am Urban, Berlin
  - Herzzentrum Brandenburg in Bernau, Bernau bei Berlin
  - CardioVascular Center Frankfurt, Frankfurt
  - Medizinisches Versorgungszentrum Prof. Mathey, Prof. Schofer GmbH, Hamburg
  - Herzzentrum Leipzig - Universitätsklinik, Leipzig
  - German Heart Center Munich, Munich
- Italy (2):
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Netherlands (2):
  - Amphia Ziekenhuis, Breda
  - University Medical Center Groningen, Groningen
- C. Hospitalar Vila Nova de Gaia/Espinho, E.P.E., Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided